CLINICAL TRIAL: NCT04686955
Title: The Efficacy of Patients With Moderate to Severe Atopic Dermatitis Treated With Chinese Herbal Medicine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-02-017A
Record Dates: First submitted 2020-12-16; First posted 2020-12-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatits; Chinese herbal medicine; Integrative medicine
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive Xiao-Xian-Gui-Fu-Tang(VGH4) for 6 weeks, then entry 2 weeks wash-out period. Then switch to receive the placebo for another 6 weeks.
  Interventions: Drug: Xiao-Xian-Gui-Fu-Tang; Drug: Placebo
- Group B (Placebo Comparator): Group B will receive placebo for 6 weeks, then entry 2 weeks wash-out period. Then switch to receive the Xiao-Xian-Gui-Fu-Tang (VGH4)for another 6 weeks.
  Interventions: Drug: Xiao-Xian-Gui-Fu-Tang; Drug: Placebo

INTERVENTIONS:
Drug: Xiao-Xian-Gui-Fu-Tang — The Xiao-Xian-Gui-Fu-Tang (VGH4) includes Xiao-Feng-San 2.0g, Dang-Gui-Yin-Zi 1.2g, Bai-Xian-Pi (Cortex Dictamni Radicis) 0.4g, and Di-Fu-Zi (Fructus Kochiae) 0.5g. The Xiao-Xian-Gui-Fu-Tang (VGH4) will be manufactured, packaged, and labeled by the KO DA Pharmaceutical Company (Taoyuan, Taiwan), under good manufacturing practice (GMP) standards.
Drug: Placebo — Matching placebo composed of inert excipients with similar color, taste, and odor, administered orally daily.

SUMMARY:
Conduct a clinical trial of integration of Chinese and Western medicine to evaluate whether the association of traditional Chinese medicine therapy has a remission effect on atopic dermatitis, and to explore the remission of lesions after an association of Chinese herbal medicine, and the correlation of syndrome differentiation types before and after treatment with Chinese and Western medicine, with a view to better understand the efficacy of atopic dermatitis in the treatment of the same disease in Traditional Chinese Medicine, and provide another option for patients with atopic dermatitis.

DETAILED DESCRIPTION:
This examination will be posted at Taipei Veterans General Hospital to recruit 24 participants who meet the inclusion criteria of atopic dermatitis to do the study. After participants agreeing to the clinical study and signing the consent form, the investigators are going to separate them into the A group (12 participants) and the B group (12 participants). The tests are going to take a total of 14 weeks.

Participants need to pass the international diagnostic criteria Hannifin and Rajka to be determined as patients with atopic dermatitis. After, participants need test by scoring Atopic Dermatitis Index (SCORAD) to be determined as mild to moderate atopic dermatitis and accept the Wang Qi Traditional Chinese Medical Constitutional Scale (TCMCS), dermatological quality of life index (DLQI) score or children's skin disease quality of life index (CDLQI) score, routine blood tests, liver and kidney function tests, immunological markers associated with atopic dermatitis Diagnosis of (eosinophils count, ECP, and IgE), tongue diagnosis, and pulse diagnosis. After the collection of data is completed, the investigators will be analyzing the data by SPSS version 21 as a two-paired t-test, ANOVA statistical method, and P <0.05 as a significant result.

ELIGIBILITY:
Inclusion Criteria:

* 6 years old to 30 years old.
* Diagnosis as an atopic dermatitis patient.
* The score of the SCORAD is over 25. (moderate to severe atopic dermatitis)

Exclusion Criteria:

* Secondary bacterial infections
* Received oral or intravenous steroid treatment, anti-biotics, phototherapy, or other immunosuppressive therapies in the previous 2 months.
* Received Chinese herbal medicine treatment or acupuncture.
* Pregnant woman or current breastfeeding.
* Who had catastrophes illness now or in the past must be avoided.
* Can not sign informed consent or can not communicate with the researcher.
* Abnormal liver enzymes.
* Abnormal kidney function tests (1.5 times higher than the upper normal limit)

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of SCORing Atopic Dermatitis(SCORAD) Index | week 0, 3, 6, 8, 11, 14
  SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). Dermatologists may use this tool before and after treatment to determine whether the treatment has been effective.
Changes of Dermatology Life Quality Index(DLQI) | week 0, 3, 6, 8, 11, 14
  The DLQI is designed to measure the health-related quality of life of adult patients suffering from a skin disease.
Changes of Children's Dermatology Life Quality Index(CDLQI) | week 0, 3, 6, 8, 11, 14
  The Children's Dermatology Life Quality Index (CDLQI) is designed to measure the impact of any skin disease on the lives of children.

SECONDARY OUTCOMES:
Blood test (AST) | week 0, 6, 14
  blood test at baseline, week 6, and follow-up (14 weeks)
Blood test (ALT) | week 0, 6, 14
  blood test at baseline, week 6, and follow-up (14 weeks)
Blood test (Serum Creatinine) | week 0, 6, 14
  blood test at baseline, week 6, and follow-up (14 weeks)
Changes of Constitution in Chinese Medicine Questionnaire | week 0, 6, 14
  The Constitution in Chinese Medicine Questionnaire (CCMQ) consists of 60 items to classify a person into one or more of nine Body constitution(BC) types: gentleness (8 Items), Qi-deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), phlegm-wetness (8 Items), wetness-heat (6 Items), blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items). Coexistence of multiple imbalanced BC types was possible which is consistent with the TCM theories. The scoring algorithm proposed in the original CCMQ was adopted in this study. A higher score in the CCMQ BC scale indicates a higher likelihood of the specific BC type, and a score of 30 is set as threshold for case definition. The CCMQ will be conducted at baseline, 12 weeks, and follow-up (16 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Pey Chen, MD, Principal Investigator — Center for Traditional Medicine, Taipei Veterans General Hospital
Locations (2):
- Taiwan (2):
  - Center for Traditional Medicine, Taipei VGH, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No